CLINICAL TRIAL: NCT06204393
Title: Effect of COVID-19 Infection on Thyroid Function and Psychological Status in Patients With Hyperthyroidism-one-year Intervention and Follow-up
Brief Title: To Investigate the Effect of 2019 Novel Coronavirus Infection on the Condition of Patients With Hyperthyroidism
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, kuanxiao Tang, chief physician, Qilu Hospital of Shandong University
Other Study IDs: KYLL-202307-049
Record Dates: First submitted 2023-12-12; First posted 2024-01-12 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2023-12

CONDITIONS: Graves Disease; COVID-19
MeSH Terms: conditions — Graves Disease; COVID-19 | interventions — Psychosocial Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- COVID-19 has a course of less than 6 days: COVID-19 is mild in hyperthyroidism patients with short course of disease.
  Interventions: Other: Thyroid metabolic index
- COVID-19 has a course of 6-9 days: The symptoms and immune level of COVD-19 in this group are in the middle level.
  Interventions: Other: Thyroid metabolic index
- COVID-19 has a course of more than 9 days: Theoretically, the symptoms and immune level of COVD-19 in this group are the worst.
  Interventions: Other: Thyroid metabolic index

INTERVENTIONS:
Other: Thyroid metabolic index — The following indicators were collected from these patients: hyperthyroidism symptoms, signs, hyperthyroidism complications, psychological evaluation results, other complications，blood routine, liver and kidney function, thyroid function (FT3, FT4, TSH), thyroid-related antibodies, glucose and lipid metabolism (FBG, HbA1c, TC, TG, HDL-C, LDL-C), thyroid ultrasound and hyperthyroidism medication.
  Psychological evaluations (using the 7-item Generalized Anxiety Disorder Questionnaire, GAD-7, and the Patient Health Questionnaire 9, PHQ-9) and interventions.
  Other Names: psychological evaluations; psychological interventions

SUMMARY:
The goal of this observational study is to learn about the correlation between COVID-19 and hyperthyroidism in Patients with hyperthyroidism complicated with COVID-19. The main questions it aims to answer are：

* The main research object is Graves disease (GD) patients.
* Changes of hyperthyroidism in GD patients complicated with COVID-19
* Changes of anxiety and depression in GD patients before and after SARS-CoV-2 infection.
* The effect of psychological intervention in GD patients after COVID-19. Participants will have regular follow-upfor one year to hyperthyroidism in our hospital, and the investigators will collect the thyroid function and related examination indexes of patients in the corresponding time period.

DETAILED DESCRIPTION:
Longitudinal analysis of GD status was performed: Three follow-up time points were identified: before COVID-19, three months and one year after recovering from COVID-19 (the first follow-up visit, the second follow-up visit. Main collection items: Hyperthyroidism symptoms, signs, hyperthyroidism complications, psychological evaluation results, other complications，blood routine, liver and kidney function, thyroid function (FT3, FT4, TSH), thyroid-related antibodies, glucose and lipid metabolism (FBG, HbA1c, TC, TG, HDL-C, LDL-C), thyroid ultrasound and hyperthyroidism medication.Through this to understand the changes of hyperthyroidism in HT patients complicated with COVID-19 and the changes of anxiety and depression in hyperthyroidism patients before and after SARS-CoV-2 infection.And the effect of psychological intervention in GD patients after COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. According to the diagnostic criteria of hyperthyroidism in the Chinese Guidelines for the Diagnosis and Treatment of Thyroid Diseases formulated by the Chinese Society of Endocrinology of the Chinese Medical Association, the patient had been diagnosed with hyperthyroidism.
2. In accordance with the diagnostic criteria of "The diagnosis and Treatment Protocol for novel coronavirus Infection (Trial version 10).

Exclusion Criteria:

1. Cases with incomplete data
2. Patients with severe autoimmune diseases, hematological diseases and malignant tumors
3. Immunodeficiency (e.g.AIDS, long-term use of corticosteroids or other immunosuppressive drugs leading to immunodeficiency)
4. Follow-up was less than 30 days
5. The results of thyroid function were less than 3 times

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cases came from HT patients who were followed up in the outpatient department of general medicine of Qilu Hospital of Shandong University, and a total of 120 hyperthyroidism patients were enrolled, who are in the maintenance stage of HT treatment and have a history of COVID-19 in the past 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-01-07 (Actual); Primary Completion 2024-08-07 (Estimated); Study Completion 2024-08-07 (Estimated)

PRIMARY OUTCOMES:
Serum TSH were measured with chemiluminescence method. | Up to 9 months
  TSH in µIU/mL
Serum FT4 were measured with chemiluminescence method. | Up to 9 months
  FT4 in pmmol/L
Serum FT3were measured with chemiluminescence method. | Up to 9 months
  FT3 in pmmol/L
Serum TRAb were measured with chemiluminescence method. | Up to 9 months
  TRAb in IU/L
Serum TPO-Ab were measured with chemiluminescence method. | Up to 9 months
  TPO-Ab in IU/ml
Serum TTG-Ab were measured with chemiluminescence method. | Up to 9 months
  TG-Ab in IU/ml
Assess the changes of patients' psychological state with Generalized Anxiety Disorder-7 Items Scale（GAD-7) | Up to 9 months
  Evaluation of anxiety state by GAD-7 scale. The lowest score of DAD-7 is 0, and the highest score is 21. The higher the score, the heavier the anxiety.
Assess the changes of patients' psychological state with Patient Health Questionnaire-9（PHQ-9） | Up to 9 months
  Evaluation of depression by PHQ-9 scale. The lowest score of PHQ-9 is 0, and the highest score is 27. The higher the score, the heavier the depression.

CONTACTS AND LOCATIONS:
Overall Officials: Kuanxiao Tang, M.D., Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided